CLINICAL TRIAL: NCT02319005
Title: A Phase 3 Multicenter, Multinational, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ALN TTRSC in Patients With Transthyretin (TTR) Mediated Familial Amyloidotic Cardiomyopathy (FAC)
Brief Title: ENDEAVOUR: Phase 3 Multicenter Study of Revusiran (ALN-TTRSC) in Patients With Transthyretin (TTR) Mediated Familial Amyloidotic Cardiomyopathy (FAC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALN-TTRSC-004
Record Dates: First submitted 2014-12-12; First posted 2014-12-18 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Transthyretin (TTR) Mediated Familial Amyloidotic Cardiomyopathy (FAC); Amyloidosis, Hereditary; Amyloid Neuropathies, Familial; Amyloid Neuropathies; Amyloidosis, Hereditary, Transthyretin-Related; Familial Transthyretin Cardiac Amyloidosis
Keywords: Cardiomyopathy; Heart Failure; FAC; Amyloid; Transthyretin; TTR; RNAi therapeutic
MeSH Terms: conditions — Amyloidosis, Familial; Amyloid Neuropathies, Familial; Amyloid Neuropathies; Amyloidosis, Hereditary, Transthyretin-Related; Cardiomyopathies; Heart Failure; Alzheimer Disease | interventions — revusiran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Revusiran (ALN-TTRSC) (Active Comparator): administered by subcutaneous (SC) injection
  Interventions: Drug: Revusiran (ALN-TTRSC)
- Sterile Normal Saline (0.9% NaCl) (Placebo Comparator): administered by subcutaneous (SC) injection
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: Revusiran (ALN-TTRSC)
  Arms: Revusiran (ALN-TTRSC)
Drug: Sterile Normal Saline (0.9% NaCl)
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of revusiran (ALN-TTRSC) in patients with transthyretin (TTR) mediated Familial Amyloidotic Cardiomyopathy. Dosing has been discontinued; patients are being followed-up for safety.

ELIGIBILITY:
Inclusion Criteria:

* Documented TTR mutation
* Amyloid deposits in cardiac or non-cardiac tissue
* Medical history of heart failure
* Evidence of cardiac involvement by echocardiogram

Exclusion Criteria:

* Has known primary amyloidosis (AL), leptomeningeal amyloidosis, non-FAC hereditary cardiomyopathy, hypertensive cardiomyopathy, or cardiomyopathy due to valvular heart disease
* Has known peripheral vascular disease affecting ambulation
* Has a Polyneuropathy Disability score >2
* Has a New York Heart Association (NYHA) classification of IV

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2014-12; Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Gollob, MD, Study Director — Alnylam Pharmaceuticals
Locations (52):
- United States (33):
  - Clinical Trial Site, Bakersfield, California
  - Clinical Trial Site, Beverly Hills, California
  - Clinical Trial Site, La Mesa, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Stanford, California
  - Clinical Trial Site, Torrance, California
  - Clinical Trial Site, Aurora, Colorado
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, New Orleans, Louisiana
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Detroit, Michigan
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, Newark, New Jersey
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Rosedale, New York
  - Clinical Trial Site, The Bronx, New York
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Cleveland, Ohio
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Charleston, South Carolina
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Fort Worth, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Richmond, Virginia
  - Clinical Trial Site, Seattle, Washington
- Belgium (3):
  - Clinical Trial Site, Anderlecht
  - Clinical Trial Site, Hasselt
  - Clinical Trial Site, Roeselare
- Clinical Trial Site, Toronto, Canada
- France (4):
  - Clinical Trial Site, Bordeaux, Aquitaine
  - Clinical Trial Site, Créteil
  - Clinical Trial Site, Marseille
  - Clinical Trial Site, Paris
- Germany (2):
  - Clinical Trial Site, Heidelberg
  - Clinical Trial Site, Münster
- Italy (3):
  - Clinical Trial Site, Bologna
  - Clinical Trial Site, Messina
  - Clinical Trial Site, Pavia
- Spain (2):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Madrid
- Clinical Trial Site, Umeå, Sweden
- United Kingdom (3):
  - Clinical Trial Site, Croydon, England
  - Clinical Trial Site, London, England
  - Clinical Trial Site, Tooting

REFERENCES:
- [Derived] Judge DP, Kristen AV, Grogan M, Maurer MS, Falk RH, Hanna M, Gillmore J, Garg P, Vaishnaw AK, Harrop J, Powell C, Karsten V, Zhang X, Sweetser MT, Vest J, Hawkins PN. Phase 3 Multicenter Study of Revusiran in Patients with Hereditary Transthyretin-Mediated (hATTR) Amyloidosis with Cardiomyopathy (ENDEAVOUR). Cardiovasc Drugs Ther. 2020 Jun;34(3):357-370. doi: 10.1007/s10557-019-06919-4. PMID 32062791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 206 patients with hereditary amyloid transthyretin (hATTR) cardiac amyloidosis were enrolled and randomized in the study.
Groups:
- Revusiran (ALN-TTRSC): All patients who received at least 1 dose of revusiran
- Placebo: All patients who received at least 1 dose of placebo
Period: Overall Study
Arm/Group | Revusiran (ALN-TTRSC) | Placebo
Started | 140 | 66
Completed | 92 | 51
Not Completed | 48 | 15

BASELINE CHARACTERISTICS:
Groups:
- Revusiran: All patients who received at least 1 dose of revusiran
- Total: Total of all reporting groups
Arm/Group | Revusiran | Placebo | Total
Number analyzed (Participants) | 140 | 66 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (9.28) | 66.2 (9.52) | 67.8 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 13 | 48
  Male | 105 | 53 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 129 | 65 | 194
  Unknown or Not Reported | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 68 | 36 | 104
  White | 66 | 29 | 95
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Distance (6-MWD)
Description: The difference between revusiran and placebo group in change from baseline to 18 months in the total distance walked in 6 minutes
Time Frame: 18 months
Population: Study drug was discontinued early due to an imbalance in mortality observed between patients treated with revusiran and placebo. No patients had an 18-month visit, therefore, the endpoints cannot be calculated as data were not collected.
Arm/Group | Revusiran | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Serum TTR Levels
Description: The difference between revusiran (ALN-TTRSC) and placebo group in the percent reduction in serum TTR levels over 18 months
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | Revusiran | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Composite Cardiovascular (CV) Mortality and Cardiovascular (CV) Hospitalization
Description: Number of cardiovascular-related deaths and cardiovascular-related hospitalizations in the placebo group compared to the revusiran (ALN-TTRSC) treatment group
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | Revusiran | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: New York Heart Association (NYHA) Class
Description: The difference between revusiran (ALN-TTRSC) and placebo group in the change from baseline to 18 months in the NYHA class
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | Revusiran | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: The difference between revusiran (ALN-TTRSC) and placebo group in the change from Baseline to 18 months in the Kansas City Cardiomyopathy Questionnaire
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | Revusiran | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Cardiovascular (CV) Mortality
Description: Number of cardiovascular-related deaths in the placebo group compared to the revusiran (ALN-TTRSC) treatment group
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | Revusiran | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Cardiovascular (CV) Hospitalization
Description: Number of cardiovascular-related hospitalizations in the placebo group compared to the revusiran (ALN-TTRSC) treatment group
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | Revusiran | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: All-cause Mortality
Description: Total number of deaths in the placebo group compared to the revusiran (ALN-TTRSC) treatment group
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | Revusiran | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) that occurred after the start of study drug administration on Day 0 (Baseline) up to 90 days post modified early termination visit (End of Study); Median duration of collection was 10 months
Description: The same event may appear as both an AE and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study
Arm/Group | Revusiran | Placebo
All-Cause Mortality (participants affected / at risk) | 23/140 | 7/66
Serious Adverse Events (participants affected / at risk) | 83/140 | 34/66
Other Adverse Events (participants affected / at risk) | 136/140 | 62/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revusiran (N=140) | Placebo (N=66)
Cardiac failure (Cardiac disorders) | 25 (35) | 9 (13)
Cardiac failure acute (Cardiac disorders) | 15 (20) | 9 (12)
Cardiac failure congestive (Cardiac disorders) | 9 (12) | 4 (6)
Atrial fibrillation (Cardiac disorders) | 7 (8) | 2 (3)
Renal failure acute (Renal and urinary disorders) | 5 (7) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 7 (7) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 3 (3)
Atrial flutter (Cardiac disorders) | 2 (2) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Cardiac failure chronic (Cardiac disorders) | 4 (4) | 2 (2)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
Renal failure (Renal and urinary disorders) | 3 (3) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 6 (6) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 2 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Subarachnoid hemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Liver function test abnormal (Investigations) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac amyloidosis (Cardiac disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nocardiosis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal amyloidosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Spleen disorders (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cutaneous Vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Lipoma excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Infective tenosynovitis (Infections and infestations) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to biliary tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumobilia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Systematic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Central nervous system lesions (Nervous system disorders) | 1 (1) | 0 (0)
Atrial Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Drug administration error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Orthostatic hypotensions (Vascular disorders) | 0 (0) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Low cardiac output syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revusiran (N=140) | Placebo (N=66)
Injection Site Pain (General disorders) | 23 (101) | 4 (13)
Injection site erythema (General disorders) | 16 (64) | 0 (0)
Fatigue (General disorders) | 14 (16) | 8 (32)
Cardiac failure (Cardiac disorders) | 10 (14) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (29) | 10 (14)
Constipation (Gastrointestinal disorders) | 20 (23) | 11 (13)
Nausea (Gastrointestinal disorders) | 20 (28) | 5 (7)
Dizziness (Nervous system disorders) | 18 (19) | 13 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (19) | 8 (9)
Neuropathy peripheral (Nervous system disorders) | 20 (21) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (22) | 9 (9)
Hypoaesthesia (Nervous system disorders) | 12 (21) | 4 (5)
Vomiting (Gastrointestinal disorders) | 9 (18) | 5 (7)
Fall (Injury, poisoning and procedural complications) | 10 (16) | 5 (9)
Atrial fibrillation (Cardiac disorders) | 16 (20) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (10) | 8 (12)
Decreased appetite (Metabolism and nutrition disorders) | 13 (16) | 6 (6)
Hypotension (Vascular disorders) | 11 (15) | 4 (4)
Gout (Metabolism and nutrition disorders) | 3 (4) | 7 (16)
Asthenia (General disorders) | 15 (18) | 2 (2)
Weight decreased (Investigations) | 12 (14) | 4 (5)
Blood lactic acid increased (Investigations) | 15 (16) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 6 (8)
Nasopharyngitis (Infections and infestations) | 11 (11) | 5 (5)
Blood bilirubin increased (Investigations) | 10 (11) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 7 (10) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 5 (5)
Bronchitis (Infections and infestations) | 10 (11) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (11) | 2 (3)
Liver function test abnormal (Investigations) | 12 (12) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (4) | 6 (9)
Sinusitis (Infections and infestations) | 7 (8) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 4 (4)
Renal failure acute (Renal and urinary disorders) | 9 (9) | 1 (3)
Fluid overload (Metabolism and nutrition disorders) | 6 (6) | 4 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 1 (1)
Insomnia (Psychiatric disorders) | 8 (8) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 9 (9) | 1 (1)

LIMITATIONS AND CAVEATS:
While dosing of patients was discontinued early, a protocol amendment allowed additional safety follow-up visits. Per the new assessment schedule, this study did not meet the criteria of a Terminated study, as additional follow-up visits occurred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT02319005/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT02319005/SAP_001.pdf